CLINICAL TRIAL: NCT03156634
Title: The Impact of the Patient Activated Learning System (PALS) on Knowledge Acquisition, Recall, and Decision Making About Antihypertensive Medication: A Pilot Study
Brief Title: A Pilot Study of the Impact of the Patient Activated Learning System (PALS) on Knowledge Acquisition, Recall, and Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1610017672
Record Dates: First submitted 2017-03-15; First posted 2017-05-17 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Patient Education
Keywords: Patient education; Internet

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view materials via one of to systems (Patient Activated Learning System or WebMD)
Who Masked: Outcomes Assessor
Masking Description: The statistician will be masked to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PALS (Experimental): Participants will view materials about the antihypertensive, chlorthalidone on the Patient Activated Learning System (PALS).
  Interventions: Other: PALS
- WedMD (Active Comparator): Participants will view materials about the antihypertensive, chlorthalidone on WebMD.
  Interventions: Other: WebMD

INTERVENTIONS:
Other: PALS — PALS is a web based patient education system that uses text and audiovisual formats to deliver patient education materials.
  Arms: PALS
Other: WebMD — WebMD is an internet based health information source.
  Arms: WedMD

SUMMARY:
This is a randomized pilot study comparing the impact of the Patient Activated Learning System (PALS) on knowledge acquisition, recall, and decision making about antihypertensive medication compared to an established online health information system (WebMD). We will also compare the two systems with regard to user experience measures such as understandability and trust.

DETAILED DESCRIPTION:
Primary research question:

1)Do hypertensive participants who learn about hypertension medication with PALS (intervention) have higher immediate and 1 week knowledge assessment scores than participants randomized to learn the same information via WebMD (control)? The investigators hypothesize that participants in the PALS group will have higher immediate and one week assessment scores.

Secondary research questions:

1. Do participants in the PALS group feel more informed to make hypothetical decisions about taking medications compared to participants in the WebMD group?

   The investigators hypothesize that participants in the PALS group will be more likely to indicate that they have sufficient information to make hypothetical decisions about taking medications than participants in the WebMD group.
2. Do participants in the PALS group rate it higher on user experience measures such as trust, usefulness, comprehensibility, and adequacy of the information, attractiveness of the site, and level of engagement, than those in the WebMD group? The investigators hypothesize ratings on these measures will be higher in the PALS group compared to the WebMD group.
3. Which questions about antihypertensives do participants consider most important and are the 5 most highly rated questions more likely to be addressed on PALS vs. WebMD? The investigators hypothesize that PALS will address more questions that participants rate as important compared to WebMD.

Participants with hypertension, who have been prescribed any antihypertensive medicine except chlorthalidone will be recruited from the Weill Cornell Internal Medicine Associates (WCIMA) practice. Potentially eligible participants who have an upcoming appointment at WCIMA will be identified via a review of the electronic medical record. In cases where the participant's eligibility is unclear, Research Assistants (RA's) will contact the participant's Primary Medical Doctor (PMD) to confirm eligibility. Potentially eligible participants will be contacted via the telephone to assess their interest in participating and to schedule a study visit for those interested. Verbal consent will be obtained either on the phone or at the study visit. Potentially eligible participants may also be recruited from the waiting room at WCIMA if the RA's were unable to contact them by phone prior to their WCIMA visit.

Eligible participants who agree to participate will be randomized to view information about the antihypertensive, chlorthalidone, via the PALS or WebMD. The study procedures will be identical for both the PALS and WebMD groups.

Chlorthalidone was chosen because, despite its efficacy, it is not prescribed as often as other antihypertensives. This will allow the investigators to select a sample of participants who are less likely to have baseline knowledge of the information we are testing.

To assess knowledge acquisition and recall, participants will be shown up to 10 pre-specified webpages within their site of randomization that contain information that answers up to 10 discrete questions about chlorthalidone. Participants will answer up to 10 corresponding assessment questions immediately after viewing the information. The knowledge score will be the percentage of correct responses. The RA's will evaluate knowledge retention by asking the same assessment questions over the phone one week later. User experience, trust, and participant decision-making will be assessed through a survey and through a short semi structured interview. The investigators will also collect information on health literacy via the REALM-SF health literacy questionnaire as well as demographic information including age, level of education, race/ethnicity, prior Internet use, and access to the Internet.

To assess question prioritization/availability on PALS/WebMD, the investigators will show participants a list of up to 40 questions and ask them to chose those most important to them. The investigators will search for the answers to the highest prioritized questions to determine availability on PALS/WebMD.

Surveys and knowledge scores will be administered via Qualtrics. Participants will be compensated with a $25 ClinCard after completing the study visit.

ELIGIBILITY:
Inclusion Criteria:

* Weill Cornell Internal Medicine Associates (WCIMA) patients with hypertension who have been prescribed any antihypertensive medicine except chlorthalidone.
* Patients who meet the criteria above and are English speaking and without cognitive impairment or other medical condition that would impair or preclude their ability to participate (such as a serious medical condition).

Exclusion Criteria:

* WCIMA patients without hypertension
* WCIMA patients with hypertension who have not been prescribed antihypertensive medicine
* Patients who are non-English speaking
* Patients with cognitive impairment or other medical condition that would impair or preclude their ability to participate (such as a serious medical condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge acquisition | Immediate
  Subjects will be asked questions about the materials they viewed.

SECONDARY OUTCOMES:
Recall | 1 week
  Subjects will be asked questions about the materials they viewed.
User experience | Immediate
  Participants will be asked about user experience including trust, usefulness, comprehensibility, and adequacy of the information, attractiveness of the site, and level of engagement of materials.
Decision making | Immediate
  Participants will be asked if they have sufficient information to make hypothetical decisions about taking chlorthalidone.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Carmel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Internal Medicine Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carmel AS, Cornelius-Schecter A, Frankel B, Jannat-Khah D, Sinha S, Pelzman F, Safford MM. Evaluation of the Patient Activated Learning System (PALS) to improve knowledge acquisition, retention, and medication decision making among hypertensive adults: Results of a pilot randomized controlled trial. Patient Educ Couns. 2019 Aug;102(8):1467-1474. doi: 10.1016/j.pec.2019.03.001. Epub 2019 Mar 4. PMID 30928344